CLINICAL TRIAL: NCT05071274
Title: A Proof of Concept Study to Evaluate the Efficacy and Tolerability of Microneedling With SkinPen in Female and Male Subjects With Facial Acne Vulgaris, Ages 18 Through 45
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crown Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-AC-21-02
Record Dates: First submitted 2021-09-22; First posted 2021-10-08 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: This proof of Concept study serves to evaluate the efficacy and tolerability of Microneedling with SkinPen in female and male Subjects with facial Acne Vulgaris, ages 18 through 45. Overall assessment of clinical outcome and safety will be based on clinic visits. The Investigator will apply an objective and precise assessment, the Lesion Count of inflammatory and non-inflammatory lesions. The Investigator will also perform the IGA assessment. Subjects will be dispensed a Diary to record any new Adverse Events between visits. Subjects will be encouraged to contact the Study Investigator if any adverse events arise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SkinPen Precision System (Experimental): After a 15-minute acclimation to ambient temperature and humidity conditions, subjects will participate in bio instrumentation to assess for erythema and will participate in standard photography.
  The Investigator will treat each subject's face from hairline to jawline with the SkinPen Precision System following instructions in the SKINPEN PRECISION SYSTEM INSTRUCTIONS with the following treatment of the face at depths of up to 1.5mm. Treatment depth will be recorded for each subject at every visit. Subjects will be dispensed a study provided diary and trained on compliance.
  Interventions: Device: Skinpen Prescision System

INTERVENTIONS:
Device: Skinpen Prescision System — Skinpen Precision is an automated nonsurgical micro needling device designed for use by licensed health care practitioners or individuals directed by practitioners. The device incorporates a sterile Microneedle cartridge and Biosheath for single use only.

SUMMARY:
This single-center, proof of concept trial is being conducted over the course of 42 days followed by a 2-month post-last treatment visit in order to assess the efficacy and tolerability of the Sponsor's SkinPen device in treating Acne Vulgaris on the face.

DETAILED DESCRIPTION:
This single-center, proof of concept trial is being conducted over the course of 42 days followed by a 2-month post-last treatment visit in order to assess the efficacy and tolerability of the Sponsor's SkinPen device in treating Acne Vulgaris on the face.

There is currently no published medical or scientific literature demonstrating the effect of Microneedling on Acne Vulgaris.

The pathogenesis of acne is attributed to four major factors:

(i)sebaceous gland hyperplasia; (ii) abnormal follicular hyperkeratinization; (iii) Propionibacterium acnes; and (iv) inflammatory and immune reactions. Increased sebum secretion is a major cause associated with the development of acne. Conventional treatments include topical retinoids, benzoyl peroxide, azelaic acid, and oral antibiotics and retinoids. However, most of these treatments take a long time to achieve a cure, and, recently, increasing resistance to antibiotics and isotretinoin's teratogenic potential have limited the use of traditional treatment.

This proof of Concept study serves to evaluate the efficacy and tolerability of Microneedling with SkinPen in female and male Subjects with facial Acne Vulgaris, ages 18 through 45. Overall assessment of clinical outcome and safety will be based on clinic visits. The Investigator will apply an objective and precise assessment, the Lesion Count of inflammatory and non-inflammatory lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females, ages 18 through 45, at the time the ICF is signed.
2. Clinical diagnosis of Acne Vulgaris
3. Investigator's Global Assessment (IGA) Score 1,2 or 3
4. Individuals willing to withhold aesthetic therapies to the areas of the face being treated or judged to potentially impact results by the Investigator (e.g. soft tissue fillers and/or any resurfacing procedures, botulinum toxin, injectable fillers, microdermabrasion, IPL (intense pulsed light), peels, facials, laser treatments, and tightening treatments, etc.) for the duration of the study. Waxing and threading is allowed but not facial laser hair removal.
5. Women of childbearing potential agree to take a urine pregnancy test at the Baseline visit. Women who are of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the baseline visit. Women must be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

   * Postmenopausal for at least 12 months prior to study;
   * Without a uterus and/or both ovaries;
   * Bilateral tubal ligation at least 6 months prior to study enrollment.
6. Individuals of childbearing potential who use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:

   1. Established use of hormonal methods of contraception (oral, injected, implanted, patch or vaginal ring) at least 3 months prior to study enrollment;
   2. Barrier methods of contraception with spermicide: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
   3. Intrauterine device (IUD) or intrauterine system (IUS)
   4. Surgical sterilization (e.g., vasectomy that has been confirmed effective by sperm count check, tubal occlusion, hysterectomy, bilateral salpingectomy/oophorectomy)
   5. Abstinence from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
7. Individuals that are willing to provide written informed consent and are able to read, speak, write and understand the informed consent document.
8. Willingness to cooperate and participate by following study requirements for the duration of the study and to report any changes in health status or medications, adverse event symptoms, or reactions immediately.

Exclusion Criteria:

1. Individuals diagnosed with known allergies to facial or general skin care products.
2. Individuals who have presence of an active systemic or local skin disease, other than Acne Vulgaris, that may affect wound healing.
3. Individuals who have severe solar elastosis.
4. Individuals with sensitivity to topical lidocaine.
5. Individuals who have physical or psychological conditions unacceptable to the Investigator.
6. Individuals who have a recent history of significant trauma to the face (< 6 months).
7. Individuals who have significant scarring, other than atrophic acne scars, in the area(s) to be treated.
8. IGA Score 0 or 4.
9. Individuals who have a recent or current history of inflammatory skin disease other than Acne Vulgaris, infection, cancerous/pre-cancerous lesion, unhealed wound in the proposed treatment areas. Individuals who have a history of systemic granulomatous diseases, active or inactive, (e.g. Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (e.g. lupus, dermatomyositis, etc.).
10. Individuals who currently have or have a history of hypertrophic scars, or keloid scars.
11. Individuals who currently have cancerous or pre-cancerous lesions in the areas to be treated and/or with a history of skin cancer.
12. Individuals who have the inability to understand instructions or to give informed consent.
13. Individuals who have had microdermabrasion or glycolic acid treatment to the treatment area(s) within 1 month prior to study participation or who will have this treatment during the study.
14. Individuals who have a history of chronic drug or alcohol abuse.
15. Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
16. Individuals who, in the Investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
17. Individuals who are current smokers or have smoked in the last 5 years.
18. Individuals who have a history of the following cosmetic treatments in the area(s) to be treated:

    * Skin tightening procedure within the past year;
    * Injectable filler of any type within the past:

      * 12 months for Hyaluronic acid fillers (e.g. Restylane)
      * 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse)
      * 24 months for Poly-L-Lactic acid fillers (e.g. Sculptra)
      * Ever for permanent fillers (e.g. Silicone, ArteFill)
    * Neurotoxins within the past 3 months;
    * Ablative resurfacing laser treatment within the past year;
    * Non-ablative, rejuvenative laser or light treatment within the past 6 months;
    * Surgical dermabrasion or deep facial peels within the past 6 months;
    * Had a chemical peel, dermabrasion, non-ablative laser or fractional laser resurfacing of the face and neck within 6 months
19. Individuals with a history of using the following prescription and over-the-counter medications:

    * Accutane or other systemic retinoids within the past 6 months;
    * Topical Retinoids or Steroids within the past 2 weeks;
    * Prescription strength skin lightening devices (e.g. hydroquinone, tretinoin, AHA, BHA and polyhydroxy acids, 4-hydroxyanisole alone or in combination with tretinoin, etc.) within 4 months;
    * Any anti-wrinkle, skin lightening devices, or any other device or topical or systemic medication known to affect skin aging or dyshcromia (devices containing alpha/beta/poly-hydroxy acids, vitamin C, soy, Q-10, hydroquinone; systemic or licorice extract (topically), Tego® Cosmo C250, gigawhite, lemon juice extract (topically), emblica extract, etc.) within 2 weeks;
    * Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use); and/or
    * Psychiatric drugs that in the Investigator's opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.
    * Topical Acne treatments including over-the-counter preparations
    * Topical anti-inflammatory agents, or
    * Topical antibiotics
20. Individuals who are nursing, pregnant, or planning to become pregnant during the study according to subject self-report.
21. Individuals having a health condition and/or pre-existing or dormant dermatologic disease, other than Acne Vulgaris, on the face or body (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
22. Individuals with a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation as determined by study documentation.
23. Individuals with an uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
24. Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures during the course of the study.
25. Individuals who are currently participating in any other study involving the use of investigational device or drugs at another research facility or doctor's office within 4 weeks prior to inclusion into the study.
26. Individuals who have observable suntan, nevi, excessive hair, etc. or other dermal conditions on the face that might influence the test results in the opinion of the Investigator or designee.
27. Individuals who have any condition, which in the opinion of the Investigator makes the patient unable to complete the study per protocol (e.g. patients not likely to avoid other facial cosmetic treatments; patients not likely to stay in the study for its duration because of other commitments, concomitant conditions, or past history; patients anticipated to be unreliable, or patients who have a concomitant condition that may develop symptoms that might confuse or confound study treatments or assessments).
28. Individuals who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
29. Subjects who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Inflammatory and Non inflammatory Lesion count | Through the course of the study, 120 days
  The primary endpoint of the study is reduction of lesion count from Visit 1 (baseline) to Visit 5, in the inflammatory (papules and pustules) and non-inflammatory (open and closed comedones) lesions.

SECONDARY OUTCOMES:
Investigators Global Assessment (IGA) | Through the course of the study, 120 days
  IGA:Score 1= almost clear, score 2 = mild severity, score 3 = moderate severity

CONTACTS AND LOCATIONS:
Locations (1):
- Crown Laboratories, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided